CLINICAL TRIAL: NCT05718011
Title: Comparison of Prophylactic Use of Dexmedetomidine and Ketamine for Prevention of Shivering After Spinal Anesthesia
Brief Title: Prevention of Shivering After Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pakistan Air Force (PAF) Hospital Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAFHIslamabad2
Record Dates: First submitted 2022-10-22; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Shivering
Keywords: Spinal anesthesia; Postoperative Shivering; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine (Experimental): 0.5 micrograms/kg
  Interventions: Drug: Dexmedetomidine
- ketamine (Active Comparator): 0.5 milligram/kg
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5 micrograms/kg diluted in 10mL of normal saline 0.9% given as IV infusion over 10 minutes
  Arms: dexmedetomidine
Drug: Ketamine — 0.5 milligrams/kg diluted in 10mL of normal saline 0.9% given as IV infusion over 10 minutes
  Arms: ketamine

SUMMARY:
Recently, ketamine and dexmedetomidine have been used to prevent shivering during anaesthesia, with good results. Ketamine (a competitive NMDA receptor antagonist) plays a role in thermoregulation at various levels and ketamine, has been shown to inhibit postoperative shivering in some reports and studies.

DETAILED DESCRIPTION:
Spinal anaesthesia is a safe and popular anaesthetic technique for various surgeries. Around 40-60% of the patients under spinal anaesthesia develop shivering.The main causes of shivering intra and postoperatively are temperature loss, decreased sympathetic tone and systemic release of pyrogens. Hypothermia during neuraxial anesthesia develops initially from core to peripheral redistribution of body heat. Redistribution of body heat during spinal or epidural anesthesia typically decreases core body temperature 0.5-1.0 degree Celsius.

Shivering is characterised by involuntary oscillatory contractions of skeletal muscles. Once the body is exposed to cold, it is a physiological response for heat preservation after peripheral vasoconstriction. Postoperative shivering is defined as the fasciculation of the face, jaw or head or muscle hyperactivity, lasting longer than 15 seconds. It is a common and challenging aspect of anaesthesia and targeted temperature modulation because it leads to increase oxygen consumption and increases the risk of hypoxia.

The most frequent complication in postoperative period is shivering which is reported to be between 20-70% after general anaesthesia. The incidence reported in previous studies are 5-65% after general anaesthesia and 30-33% after epidural procedures. The overall shivering incidence in a recent meta-analysis was 34%.

The underlying pathology of shivering is not fully understood yet, therefore the definitive treatment and prevention has not been established till date. Due to its importance as postoperative complication and the lack of available data about aetiology and treatment, this narrative review of the published literature on this topic is essential.

Various pharmacological agents being used for prophylaxis and treatment of post spinal shivering are Opioids like fentanyl, tramadol, pethidine, Anticholinergics like physostigmine, NMDA receptor antagonist like ketamine and the latest being alpha-2 antagonists like clonidine, dexmedetomidine.

Recently, ketamine and dexmedetomidine have been used to prevent shivering during anaesthesia, with good results. Ketamine (a competitive NMDA receptor antagonist) plays a role in thermoregulation at various levels and ketamine, has been shown to inhibit postoperative shivering in some reports and studies.

Dexmedetomidine, a centrally acting alpha 2-adrenergic agonist, has been used as a sedative agent and is known to reduce the shivering threshold. Dexmedetomidine also provided sedation which is sufficient to prevent the anxiety without any adverse effects. And until date, there are limited studies using dexmedetomidine in the treatment of postoperative shivering.

A very limited data is available on this subject in our Pakistani population. Pethidine is drug of choice for the prevention and treatment of shivering. Due to the non-availability of Pethidine, doctors are looking for newer and better options. Considering this, a study is designed to compare between Dexmedetomidine and Ketamine, as they are easily available and very few studies are done till date comparing them, as ketamine isn't researched much as an anti-shivering agent as it is known for undesirable side effects like delirium and hallucinations and dexmedetomidine being a newer agent. Results of this study will help to select the better prophylactic option for prevention of shivering after spinal anaesthesia in our general population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-50 years.
* Both genders
* ASA physical status I and II
* Undergoing lower abdominal or lower limb surgeries under spinal anaesthesia

Exclusion Criteria:

* Patients with history of thyroid and neuromuscular diseases
* Patients with severe hypovolemia
* Patients with febrile illness
* Patients who required blood transfusion during surgery
* Patients with body temperature ≤ 36˚C or ≥ 38˚C on thermometer

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Postoperative Shivering | Change in every 10 minutes after spinal anesthesia till PACU discharge after 01 hour PACU stay.
  Visible muscle activity in more than one muscle group.

CONTACTS AND LOCATIONS:
Overall Officials: ATIYA CHAUDHRY, MBBS, Principal Investigator — PAF Hospital Islamabad
Locations (1):
- PAF Hospital Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bindu B, Bindra A, Rath G. Temperature management under general anesthesia: Compulsion or option. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):306-316. doi: 10.4103/joacp.JOACP_334_16. PMID 29109627
- [Background] Hoshijima H, Takeuchi R, Kuratani N, Nishizawa S, Denawa Y, Shiga T, Nagasaka H. Incidence of postoperative shivering comparing remifentanil with other opioids: a meta-analysis. J Clin Anesth. 2016 Aug;32:300-12. doi: 10.1016/j.jclinane.2015.08.017. Epub 2015 Oct 1. PMID 26432635
- [Background] Choi KE, Park B, Moheet AM, Rosen A, Lahiri S, Rosengart A. Systematic Quality Assessment of Published Antishivering Protocols. Anesth Analg. 2017 May;124(5):1539-1546. doi: 10.1213/ANE.0000000000001571. PMID 27622717
- [Background] Park SM, Mangat HS, Berger K, Rosengart AJ. Efficacy spectrum of antishivering medications: meta-analysis of randomized controlled trials. Crit Care Med. 2012 Nov;40(11):3070-82. doi: 10.1097/CCM.0b013e31825b931e. PMID 22890247
- [Background] Leite MA, Orsini M, de Freitas MR, Pereira JS, Gobbi FH, Bastos VH, de Castro Machado D, Machado S, Arrias-Carrion O, de Souza JA, Oliveira AB. Another Perspective on Fasciculations: When is it not Caused by the Classic form of Amyotrophic Lateral Sclerosis or Progressive Spinal Atrophy? Neurol Int. 2014 Aug 8;6(3):5208. doi: 10.4081/ni.2014.5208. eCollection 2014 Aug 5. PMID 25309711
- [Background] Buggy DJ, Crossley AW. Thermoregulation, mild perioperative hypothermia and postanaesthetic shivering. Br J Anaesth. 2000 May;84(5):615-28. doi: 10.1093/bja/84.5.615. No abstract available. PMID 10844839
- [Background] Bozgeyik S, Mizrak A, Kilic E, Yendi F, Ugur BK. The effects of preemptive tramadol and dexmedetomidine on shivering during arthroscopy. Saudi J Anaesth. 2014 Apr;8(2):238-43. doi: 10.4103/1658-354X.130729. PMID 24843340
- [Background] Lakhe G, Adhikari KM, Khatri K, Maharjan A, Bajracharya A, Khanal H. Prevention of Shivering during Spinal Anesthesia: Comparison between Tramadol, Ketamine and Ondansetron. JNMA J Nepal Med Assoc. 2017 Oct-Dec;56(208):395-400. PMID 29453468
- [Result] Ameta N, Jacob M, Hasnain S, Ramesh G. Comparison of prophylactic use of ketamine, tramadol, and dexmedetomidine for prevention of shivering after spinal anesthesia. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):352-356. doi: 10.4103/joacp.JOACP_211_16. PMID 30386019